CLINICAL TRIAL: NCT04516018
Title: The Effect of Prolonged Shivering Thermogenesis on Glucose Homeostasis in Overweight/Obese Humans
Brief Title: Shivering and Glucose Homeostasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL73487.068.20
Record Dates: First submitted 2020-07-24; First posted 2020-08-17 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Healthy Overweight/Obese
Keywords: Type 2 diabetes mellitus; Shivering thermogenesis; skeletal muscle
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: a single arm, longitudinal study (10-day intermittent shivering exposure) in a pre-post design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cold acclimation arm (Experimental): An oral glucose tolerance test will be performed on day 1 of the study. The next day (day 2), subjects will be exposed to shivering thermogenesis for at least 1 hour. The day after, an oral glucose tolerance test will be performed (day 3). The following 9 days, subjects will be exposed daily to shivering thermogenesis for at least 1 hour (day 4-12). On the last day (day 13), an oral glucose tolerance test will be performed.
  Interventions: Other: Cold exposure

INTERVENTIONS:
Other: Cold exposure — Subjects will be exposed to shivering thermogenesis for at least 1 hour for 10 days

SUMMARY:
The purpose of this study is to investigate the effect of prolonged shivering thermogenesis on glucose homeostasis in overweight/obese humans.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Caucasian
* Healthy (as determined by dependent physician based on medical questionnaire)
* Man, or postmenopausal (defined as at least 1year post cessation of menses) woman
* Aged 40 - 75 years at the start of the study
* BMI 27 and 35 kg/m2
* Stable dietary habits (no weight loss or gain >3kg in the past 3 months)

Exclusion Criteria:

* - Not meeting all inclusion criteria
* Medication use known to hamper subject's safety during study procedures
* Co-morbidities to which the intervention or program that may pose as a complicating factor
* Subjects diagnosed with cardiovascular diseases or cancer
* Fasting plasma glucose ≥ 7.0 mmol/l
* Haemoglobin < 7.8 mmol/l for women, or < 8.4 mmol/l for men
* Previously diagnosed with type 2 diabetes
* Abuse alcohol/drug abuse
* Subjects who do not want to be informed about unexpected medical findings during the screening/study or do not wish that their physician is informed.
* Engagement in structured exercise > 2h per week
* Participation in another biomedical study within 1 month before the first study
* Smoking
* Cold-acclimated, such as takes daily extended cold baths, works in a refrigerated environment, or regular cold-water swimming within 1 month of starting the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
area under the curve (AUC) of the glucose tolerance test | 1 day following cold exposure and following 9 consecutive days of cold exposure
  area under the curve (AUC) of the glucose tolerance test before cold exposure, 1 day after cold exposure and after 9 consecutive days of cold exposure.

SECONDARY OUTCOMES:
skeletal muscle GLUT4 translocation | 1 day following cold exposure and following 9 consecutive days of cold exposure
  Comparison between skeletal muscle GLUT4 translocation, as assessed by wide-field microscopy both before and after cold acclimation

OTHER OUTCOMES:
Insulin sensitivity | 1 day following cold exposure and following 9 consecutive days of cold exposure
  Comparison between insulin sensitivity as estimated from the insulin and glucose concentrations during the OGTT both before and after cold acclimation.
Heart rate | 1 day following cold exposure and following 9 consecutive days of cold exposure
  Comparison between heart rate during cold exposure both before and after cold acclimation
Blood pressure | 1 day following cold exposure and following 9 consecutive days of cold exposure
  Comparison between blood pressure during cold exposure both before and after cold acclimation
Energy expenditure | 1 day following cold exposure and following 9 consecutive days of cold exposure
  Comparison between energy expenditure as assessed by indirect calorimetry both before and after cold acclimation
Substrate oxidation | 1 day following cold exposure and following 9 consecutive days of cold exposure
  Comparison between substrate oxidation as assessed by indirect calorimetry both before and after cold acclimation
Plasma substrates | 1 day following cold exposure and following 9 consecutive days of cold exposure
  Comparison between plasma substrates change during cold acclimation (including insulin, FFA, glucose) both before and after cold acclimation
Plasma hormones | 1 day following cold exposure and following 9 consecutive days of cold exposure
  Comparison between plasma hormones change during cold acclimation (including insulin, FFA, glucose) both before and after cold acclimation
Skeletal muscle intramyocellular substrate content | 1 day following cold exposure and following 9 consecutive days of cold exposure
  Comparison between skeletal muscle intramyocellular substrate content both before and after cold acclimation
Protein expression in skeletal muscle | 1 day following cold exposure and following 9 consecutive days of cold exposure
  Comparison between protein expression in skeletal muscle both before and after cold acclimation of specific pathways as determined by western blot
Gene expression in skeletal muscle | 1 day following cold exposure and following 9 consecutive days of cold exposure
  Comparison between gene expression in skeletal muscle both before and after cold acclimation of specific pathways as determined by RT-qPCR
Body temperatures | 1 day following cold exposure and following 9 consecutive days of cold exposure
  Change in both skin and core temperature upon cold acclimation as assessed by means of temperatures sensors and a core temperature pill
Shivering activity | 1 day following cold exposure and following 9 consecutive days of cold exposure
  Muscle shivering activity as determined by EMG. Comparison between shivering activity before and after cold acclimation

CONTACTS AND LOCATIONS:
Overall Officials: Wouter van Marken Lichtenbelt, Prof., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Sellers AJ, van Beek SMM, Hashim D, Baak R, Pallubinsky H, Moonen-Kornips E, Schaart G, Gemmink A, Jorgensen JA, van de Weijer T, Kalkhoven E, Hooiveld GJ, Kersten S, Hesselink MKC, Schrauwen P, Hoeks J, van Marken Lichtenbelt WD. Cold acclimation with shivering improves metabolic health in adults with overweight or obesity. Nat Metab. 2024 Dec;6(12):2246-2253. doi: 10.1038/s42255-024-01172-y. Epub 2024 Dec 6. PMID 39643644